CLINICAL TRIAL: NCT00818610
Title: Beta-lactam Monotherapy Versus Beta-lactam - Macrolide Association as Empiric Antibiotherapy Strategies in Non-severe Hospitalized Community-acquired Pneumonia: a Randomized, Non-inferiority, Open Trial.
Brief Title: Monotherapy Versus Bitherapy in Non-severe Hospitalized Community-acquired Pneumonia
Acronym: BICAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss National Fund for Scientific Research (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Garin Nicolas, Associate physician, Swiss National Fund for Scientific Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3200B0-120074/1
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired infections; Pneumonia; Clinical Stability; Antibiotics; Combination therapy; Atypical bacteria
MeSH Terms: conditions — Community-Acquired Pneumonia; Community-Acquired Infections; Pneumonia | interventions — beta-Lactams; Amoxicillin; Cefuroxime; Amoxicillin-Potassium Clavulanate Combination; Macrolides; Clarithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy (Experimental)
  Interventions: Drug: Beta lactam (amoxicillin / clav. acid OR cefuroxime)
- Bi-therapy (Active Comparator)
  Interventions: Drug: Beta-lactam (amoxicillin / clav. acid OR cefuroxime) AND macrolide (clarithromycin)

INTERVENTIONS:
Drug: Beta lactam (amoxicillin / clav. acid OR cefuroxime) — 1.2 g 4x/d OR 1.5 g 3x/d IV
  Other Names: Augmentin; Zinacef
  Arms: Monotherapy
Drug: Beta-lactam (amoxicillin / clav. acid OR cefuroxime) AND macrolide (clarithromycin) — 1.2 g 4x/d OR 1.5 g 3x/d IV AND 0.5 g 2x/d IV/PO
  Other Names: Augmentin; Zinacef; Klacid
  Arms: Bi-therapy

SUMMARY:
The purpose of this study is to determine whether a monotherapy with a Beta-Lactam is not inferior to an association of a Beta-Lactam and a macrolide in treating adult patients with community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* New infiltrate on chest X-ray, unexplained by another disease process
* Presence of at least two of the following findings suggestive of pneumonia: fever or hypothermia, new or increasing cough, sputum production, pleuritic chest pain, tachypnea, dyspnea or focal signs on chest examination
* Need for hospitalization as defined by the emergency physician in charge of the patient

Exclusion Criteria:

* Allergy to one of the study drugs
* Pregnancy
* Severe immunosuppression
* Recent (<14 d) hospitalization, or currently hospitalized since > 48 hours
* Residency in a nursing home
* Previous use of more than 24 hours of any antibiotic
* Severe community-acquired pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Stability (hours) | 30 days

SECONDARY OUTCOMES:
All cause mortality | in-hospital, at 30 and at 90 days
length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Perrier, MD, Principal Investigator — University of Geneva and University Hospital of Geneva
Locations (6):
- Switzerland (6):
  - HFR-Fribourg, Hôpital Cantonal, Fribourg, Canton of Fribourg
  - Stadtspital Triemli, Zurich, Canton of Zurich
  - Centre Hospitalier du Centre du Valais, Sion, Valais
  - Hôpitaux Universitaires de Genève, Geneva
  - Hôpital Neuchâtelois - La Chaux-de-Fonds, La Chaux-de-Fonds
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Derived] Chauffard A, Bridevaux PO, Carballo S, Prendki V, Reny JL, Stirnemann J, Garin N. Accuracy of a score predicting the presence of an atypical pathogen in hospitalized patients with moderately severe community-acquired pneumonia. BMC Infect Dis. 2022 May 3;22(1):424. doi: 10.1186/s12879-022-07423-1. PMID 35505308
- [Derived] Garin N, Genne D, Carballo S, Chuard C, Eich G, Hugli O, Lamy O, Nendaz M, Petignat PA, Perneger T, Rutschmann O, Seravalli L, Harbarth S, Perrier A. beta-Lactam monotherapy vs beta-lactam-macrolide combination treatment in moderately severe community-acquired pneumonia: a randomized noninferiority trial. JAMA Intern Med. 2014 Dec;174(12):1894-901. doi: 10.1001/jamainternmed.2014.4887. PMID 25286173